CLINICAL TRIAL: NCT03917784
Title: Effect of Oral Supplementation With Curcumin on Insulin Sensitivity in Subjects With Prediabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, César Leonardo González Aguilar, Internal Medicine Resident, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DI/18/111/03/067
Record Dates: First submitted 2019-04-07; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: PreDiabetes
Keywords: Curcumin; Insulin sensitivity; HOMA
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Curcumin; Starch

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin and bioperine (Experimental): This group will receive curcumin 500 mg and bioperine 5 mg oral dosing every 12 hours for 3 months
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): This group will receive placebo (starch) 500 mg oral dosing every 12 hours for 3 months
  Interventions: Drug: Starch

INTERVENTIONS:
Drug: Curcumin — Oral supplementation with curcumin 500 mg oral dosing for 3 months
  Arms: Curcumin and bioperine
Drug: Starch — Oral supplementation with starch 500 mg oral dosing for 3 months
  Arms: Placebo

SUMMARY:
This study evaluates the effects of oral supplementation with curcumin on the insulin sensitivity in subjects with prediabetes. The half of participants will receive curcumin and bioperine in combination, while the other half receive placebo.

DETAILED DESCRIPTION:
The therapeutic strategies for prediabetes to this day are based on the change of habits, mainly food and exercise plans. It has been advice, in specific circumstances, to grant a pharmacological regimen.

Curcumin or Curcuma Longa ((1E,6E)21,7-bis(4-hydroxy-3-methoxyphenyl)-1,6- heptadiene-3,5-dione), is the main ingredient of the Hindu condiment, Turmeric, which is obtained from the Rhizome plant. In new studies, it has been documented that the oral consumption of curcumin (Curcuma longa) in pre-diabetic and diabetic patients has a positive effect as an antidiabetic agent thanks to its anti-inflammatory, antioxidant, antithrombotic, cardio and neuroprotective effects. In animal models, it has been shown that oral curcumin consumption is capable of increasing insulin sensitivity in liver, muscle and adipose tissue, increases glucose uptake in muscle and insulin secretion, which is reflected in the reduction of hyperglycemia, glycosylated hemoglobin, decrease of the homeostatic model assessment of insulin resistance (HOMA-IR) and decrease of serum lipids.

Curcumin has been included in the oriental diet since ancient times and is used in traditional medicine, which is why it is considered safe, since its consumption is approved by the FDA (Federal Drugs Administration). A 12g per day dose has shown no side effects in humans. Therefore, it is proposed that the consumption of curcumin in pre-diabetic patients can improve glucose tolerance and decrease insulin resistance parameters.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with age between 18 and 60 years old.
* With prediabetes diagnosis, according to the American Diabetes Association :

  1. Fasting serum glucose: 100-125 mg/dL
  2. Glycosylated hemoglobin (HbA1c): 5.7-6.4%
  3. Post-prandial glucose: 140-199 mg/dL after an oral dose of 75 g of glucose.

Exclusion Criteria:

* Subjects with any type of diabetes.
* Subjects with body mass index > 35 kg/m2
* Pregnant Women.
* Volunteers who ingest drugs that alter blood glucose levels, antiplatelet agents, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, fibrates, statins.
* Subjects with serum creatinine > 2 mg/dL or in renal replacement therapy.
* Subjects that normally consume food supplements.
* Subjects with acute infections or with chronical diseases (cancer, rheumatoid arthritis, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
HOMA- IR | 3 months
  (Insulin µU/ml)(Glucose mg/dl)/405.
HOMA- Beta | 3 months
  (20)(FPI)/(FPG - 3.5)
Matsuda index | 3 months
  10,000/√[(basal glucose)(basal insulin)*(glucose)(insulin)]

SECONDARY OUTCOMES:
weight | 6 weeks and 12 weeks
  weight in kilograms
height | 6 weeks and 12 weeks
  height in centimetres
waist circumference | 6 weeks and 12 weeks
  waist circumference in centimetres
hip circumference. | 6 weeks and 12 weeks
  hip circumference in centimetres
insulin | 6 weeks and 12 weeks
  insulin in µU/ml
triglycerides | 6 weeks and 12 weeks
  triglycerides in mg/dl
cholesterol | 6 weeks and 12 weeks
  cholesterol in mg/dl
HDL cholesterol | 6 weeks and 12 weeks
  HDL cholesterol in mg/dl
LDL cholesterol | 6 weeks and 12 weeks
  LDL cholesterol in mg/dl
uric acid | 6 weeks and 12 weeks
  uric acid in mg/dl
creatinine | 6 weeks and 12 weeks
  creatinine in mg/dl
urea | 6 weeks and 12 weeks
  urea in mg/dl
alanine amino transferase | 6 weeks and 12 weeks
  alanine amino transferase in U/L
alkaline phosphatase | 6 weeks and 12 weeks
  alkaline phosphatase in U/L
lactic dehydrogenase | 6 weeks and 12 weeks
  lactic dehydrogenase in U/L
glycosylated hemoglobin | 6 weeks and 12 weeks
  glycosylated hemoglobin in percentage
total bilirubin | 6 weeks and 12 weeks
  total bilirubin in mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de México Dr. Eduardo Liceaga, Mexico City, Cuauhtémoc, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Identified individual participant data for all primary and secondary outcomes measures will be made avaliable
Supporting Information: Study Protocol
Time Frame: Data will be avaliable whithin 6 months of study completion

REFERENCES:
- [Background] American Diabetes Association. 5. Prevention or Delay of Type 2 Diabetes: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S51-S54. doi: 10.2337/dc18-S005. PMID 29222376
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S13-S27. doi: 10.2337/dc18-S002. PMID 29222373
- [Background] Alibasic E, Ramic E, Alic A. Prevention of diabetes in family medicine. Mater Sociomed. 2013;25(2):80-2. doi: 10.5455/msm.2013.25.80-82. PMID 24082827
- [Background] Ferrannini E. Definition of intervention points in prediabetes. Lancet Diabetes Endocrinol. 2014 Aug;2(8):667-75. doi: 10.1016/S2213-8587(13)70175-X. Epub 2014 Jan 28. PMID 24731662
- [Result] Rojas-Martinez R, Basto-Abreu A, Aguilar-Salinas CA, Zarate-Rojas E, Villalpando S, Barrientos-Gutierrez T. [Prevalence of previously diagnosed diabetes mellitus in Mexico.]. Salud Publica Mex. 2018 May-Jun;60(3):224-232. doi: 10.21149/8566. Spanish. PMID 29746739
- [Result] Defronzo RA, Tripathy D, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Kitabchi AE, Mudaliar S, Ratner RE, Stentz FB, Musi N, Reaven PD, Gastaldelli A; ACT NOW Study. Prediction of diabetes based on baseline metabolic characteristics in individuals at high risk. Diabetes Care. 2013 Nov;36(11):3607-12. doi: 10.2337/dc13-0520. Epub 2013 Sep 23. PMID 24062330
- [Result] Abdul-Ghani MA, Abdul-Ghani T, Stern MP, Karavic J, Tuomi T, Bo I, Defronzo RA, Groop L. Two-step approach for the prediction of future type 2 diabetes risk. Diabetes Care. 2011 Sep;34(9):2108-12. doi: 10.2337/dc10-2201. Epub 2011 Jul 25. PMID 21788628
- [Result] Lamy A, Tong W, Jung H, Gafni A, Singh K, Tyrwhitt J, Yusuf S, Gerstein HC; ORIGIN Investigators. Cost implications of the use of basal insulin glargine in people with early dysglycemia: the ORIGIN trial. J Diabetes Complications. 2014 Jul-Aug;28(4):553-8. doi: 10.1016/j.jdiacomp.2014.02.012. Epub 2014 Mar 2. PMID 24684774
- [Result] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Result] Bonora E, Targher G, Alberiche M, Bonadonna RC, Saggiani F, Zenere MB, Monauni T, Muggeo M. Homeostasis model assessment closely mirrors the glucose clamp technique in the assessment of insulin sensitivity: studies in subjects with various degrees of glucose tolerance and insulin sensitivity. Diabetes Care. 2000 Jan;23(1):57-63. doi: 10.2337/diacare.23.1.57. PMID 10857969
- [Result] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Result] Chuengsamarn S, Rattanamongkolgul S, Luechapudiporn R, Phisalaphong C, Jirawatnotai S. Curcumin extract for prevention of type 2 diabetes. Diabetes Care. 2012 Nov;35(11):2121-7. doi: 10.2337/dc12-0116. Epub 2012 Jul 6. PMID 22773702
- [Result] Na LX, Li Y, Pan HZ, Zhou XL, Sun DJ, Meng M, Li XX, Sun CH. Curcuminoids exert glucose-lowering effect in type 2 diabetes by decreasing serum free fatty acids: a double-blind, placebo-controlled trial. Mol Nutr Food Res. 2013 Sep;57(9):1569-77. doi: 10.1002/mnfr.201200131. Epub 2012 Aug 29. PMID 22930403
- [Result] Chuengsamarn S, Rattanamongkolgul S, Phonrat B, Tungtrongchitr R, Jirawatnotai S. Reduction of atherogenic risk in patients with type 2 diabetes by curcuminoid extract: a randomized controlled trial. J Nutr Biochem. 2014 Feb;25(2):144-50. doi: 10.1016/j.jnutbio.2013.09.013. Epub 2013 Nov 6. PMID 24445038
- [Result] Zhao SG, Li Q, Liu ZX, Wang JJ, Wang XX, Qin M, Wen QS. Curcumin attenuates insulin resistance in hepatocytes by inducing Nrf2 nuclear translocation. Hepatogastroenterology. 2011 Nov-Dec;58(112):2106-11. doi: 10.5754/hge11219. PMID 22024084
- [Result] Kang C, Kim E. Synergistic effect of curcumin and insulin on muscle cell glucose metabolism. Food Chem Toxicol. 2010 Aug-Sep;48(8-9):2366-73. doi: 10.1016/j.fct.2010.05.073. Epub 2010 Jun 1. PMID 20561944
- [Result] Shao W, Yu Z, Chiang Y, Yang Y, Chai T, Foltz W, Lu H, Fantus IG, Jin T. Curcumin prevents high fat diet induced insulin resistance and obesity via attenuating lipogenesis in liver and inflammatory pathway in adipocytes. PLoS One. 2012;7(1):e28784. doi: 10.1371/journal.pone.0028784. Epub 2012 Jan 9. PMID 22253696
- [Result] Abdel Aziz MT, El-Asmar MF, El Nadi EG, Wassef MA, Ahmed HH, Rashed LA, Obaia EM, Sabry D, Hassouna AA, Abdel Aziz AT. The effect of curcumin on insulin release in rat-isolated pancreatic islets. Angiology. 2010 Aug;61(6):557-66. doi: 10.1177/0003319709356424. Epub 2010 Apr 14. PMID 20395228
- [Result] Aziz MT, El-Asmar MF, Rezq AM, Wassef MA, Fouad H, Roshdy NK, Ahmed HH, Rashed LA, Sabry D, Taha FM, Hassouna A. Effects of a novel curcumin derivative on insulin synthesis and secretion in streptozotocin-treated rat pancreatic islets in vitro. Chin Med. 2014 Jan 14;9(1):3. doi: 10.1186/1749-8546-9-3. PMID 24422903
- [Result] Hu GX, Lin H, Lian QQ, Zhou SH, Guo J, Zhou HY, Chu Y, Ge RS. Curcumin as a potent and selective inhibitor of 11beta-hydroxysteroid dehydrogenase 1: improving lipid profiles in high-fat-diet-treated rats. PLoS One. 2013;8(3):e49976. doi: 10.1371/journal.pone.0049976. Epub 2013 Mar 22. PMID 23533564
- [Result] Nagabhushan M, Bhide SV. Curcumin as an inhibitor of cancer. J Am Coll Nutr. 1992 Apr;11(2):192-8. PMID 1578097
- [Result] Azuine MA, Bhide SV. Chemopreventive effect of turmeric against stomach and skin tumors induced by chemical carcinogens in Swiss mice. Nutr Cancer. 1992;17(1):77-83. doi: 10.1080/01635589209514174. PMID 1574446
- [Result] Huang MT, Lou YR, Ma W, Newmark HL, Reuhl KR, Conney AH. Inhibitory effects of dietary curcumin on forestomach, duodenal, and colon carcinogenesis in mice. Cancer Res. 1994 Nov 15;54(22):5841-7. PMID 7954412
- [Result] Mohammadi A, Sahebkar A, Iranshahi M, Amini M, Khojasteh R, Ghayour-Mobarhan M, Ferns GA. Effects of supplementation with curcuminoids on dyslipidemia in obese patients: a randomized crossover trial. Phytother Res. 2013 Mar;27(3):374-9. doi: 10.1002/ptr.4715. Epub 2012 May 21. PMID 22610853
- [Result] Ganjali S, Sahebkar A, Mahdipour E, Jamialahmadi K, Torabi S, Akhlaghi S, Ferns G, Parizadeh SM, Ghayour-Mobarhan M. Investigation of the effects of curcumin on serum cytokines in obese individuals: a randomized controlled trial. ScientificWorldJournal. 2014 Feb 11;2014:898361. doi: 10.1155/2014/898361. eCollection 2014. PMID 24678280

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03917784/Prot_SAP_000.pdf